CLINICAL TRIAL: NCT01481441
Title: Quantification of Contrast Enhanced Ultrasound (CEUS) in the Detection of Prostate Cancer
Acronym: AMC_2011_190
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: New study protocol started including targeted biopsies
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. dr. ir. H. Wijkstra, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL37231.018.11
Record Dates: First submitted 2011-11-21; First posted 2011-11-29 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: Contrast Enhanced Ultrasound (CEUS); Prostate cancer; Quantification; Prostate biopsies; Transrectal ultrasound (TRUS); Microbubbles
MeSH Terms: conditions — Prostatic Neoplasms | interventions — contrast agent BR1; Powders; Solvents; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SonoVue (Other): Ultrasound Contrast Agent
  Interventions: Drug: SonoVue

INTERVENTIONS:
Drug: SonoVue — 2.4 ml Bolus Injection by intravenous canule. Multi-repeatable (up to 4 bolus) if necessary.
  Other Names: SonoVue sulphur hexafluoride microbubbles 8 microlitres/ml; Powder and solvent for dispersion for injection.; MARKETING AUTHORISATION NUMBER(S): EU/1/01/177/002

SUMMARY:
With Contrast Enhanced UltraSound (CEUS) cancer induced neovascularisation can be visualised with the potential to improve ultrasound imaging for prostate cancer detection and localisation significantly. The past years numerous studies have been performed with CEUS, all basing their results on subjective judgement of the investigator. CEUS image interpretation is difficult and requires a well-trained expert. To overcome these difficulties CEUS quantification techniques can be of use. The techniques used in this protocol have been developed in cooperation with the Technical University in Eindhoven (TU/e) and BRACCO, Geneva.

The investigators hypothesize improvement of the PCa detection rate with quantification, compared with subjective CEUS interpretation and known numbers in literature.

Also a comparison between quantification results and tumour differentiation grade (Gleason score) will be made, the investigators hypothesize a positive correlation.

ELIGIBILITY:
Population:

All patients already scheduled for biopsy because of a raised Prostate-Specific Antigen (PSA) and/ or abnormal Digital Rectal Examination (DRE) in the Academic Medical Centre (AMC), excluding patients who do meet the exclusion criteria.

Inclusion criteria:

* age ≥ 18 years
* signed informed consent

Exclusion criteria:

* Has documented acute prostatitis or urinary tract infections.
* History of any clinically unstable cardiac condition including class III/IV cardiac failure or right-to-left shunts.
* Has had severe cardiac rhythm disorders within the last 7 days.
* Has severe pulmonary hypertension (pulmonary artery pressure >90 mmHg) or uncontrolled systemic hypertension or respiratory distress syndrome
* Has received a biopsy procedure within 30 days before admission into this study
* Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study.
* Is incapable of understanding the language in which the information for the patient is given.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2011-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Quantification prediction compared with prostate biopsy histology | 3 years
  Prostate cancer detection rate by quantification.
  Answering the question: What is the difference in, for malignancy suspicious, areas between CEUS quantification and subjective interpretation in relation to the histological biopsy results?

SECONDARY OUTCOMES:
Quantification prediction compared with prostate biopsy histology | 3 years
  Prostate cancer Gleason score compared to quantification results
  Answering the question: Is there a relation between Gleason score and quantification results?

CONTACTS AND LOCATIONS:
Overall Officials: H. Wijkstra, Prof. Dr. Ir., Principal Investigator — AMC University Hospital
Locations (1):
- AMC University Hospital, Amsterdam, Netherlands

REFERENCES:
- [Result] Postema AW, Frinking PJ, Smeenge M, De Reijke TM, De la Rosette JJ, Tranquart F, Wijkstra H. Dynamic contrast-enhanced ultrasound parametric imaging for the detection of prostate cancer. BJU Int. 2016 Apr;117(4):598-603. doi: 10.1111/bju.13116. Epub 2015 Jun 29. PMID 25754526